CLINICAL TRIAL: NCT02573922
Title: Opioid Induced Bowel Dysfunction in Patients Undergoing Spinal Surgery
Acronym: oksineukir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Merja Kokki, MD, PhD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH24-02-2012
Record Dates: First submitted 2015-10-09; First posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Constipation
Keywords: constipation; opioid; Oxycodone; Oxycodone-naloxone; spine surgery
MeSH Terms: conditions — Constipation | interventions — oxycodone naloxone combination; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodone-naloxone (Experimental): Oxycodone-naloxone prolonged release tablet twice a day
  Interventions: Drug: oxycodone-naloxone
- Oxycodone (Active Comparator): Oxycodone prolonged release tablet twice a day
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: oxycodone-naloxone
  Arms: Oxycodone-naloxone
Drug: Oxycodone
  Arms: Oxycodone

SUMMARY:
In the present study, the primary aim was to evaluate if oxycodone-naloxone combination compared to oxycodone reduced opioid induced constipation in patients with or without chronic opioid treatment undergoing spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* BMI 17 - 35 kg/m2
* elective spine surgery
* informed consent obtained

Exclusion Criteria:

* allergy to the used drugs
* other contraindication to oxycodone medication
* no informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
opioid induced constipation | from the surgery up to 21 days
  Opioid induced constipation was assessed with bowel function index

CONTACTS AND LOCATIONS:
Overall Officials: Merja Kokki, MD, PhD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

REFERENCES:
- [Derived] Kuronen M, Kokki H, Nyyssonen T, Savolainen S, Kokki M. Life satisfaction and pain interference in spine surgery patients before and after surgery: comparison between on-opioid and opioid-naive patients. Qual Life Res. 2018 Nov;27(11):3013-3020. doi: 10.1007/s11136-018-1961-x. Epub 2018 Aug 2. PMID 30073471
- [Derived] Kokki M, Kuronen M, Naaranlahti T, Nyyssonen T, Pikkarainen I, Savolainen S, Kokki H. Opioid-Induced Bowel Dysfunction in Patients Undergoing Spine Surgery: Comparison of Oxycodone and Oxycodone-Naloxone Treatment. Adv Ther. 2017 Jan;34(1):236-251. doi: 10.1007/s12325-016-0456-9. Epub 2016 Dec 5. PMID 27921252